CLINICAL TRIAL: NCT01946087
Title: Remote Ischemic Preconditioning Induces Myocardial RISK Signaling Pathway in Patients Undergoing Valvular Heart Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2012-0283
Record Dates: First submitted 2013-09-04; First posted 2013-09-19 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Patients With Elective Aortic Valve Replacement
Keywords: Remote ischemic preconditioning; cardiac surgery; left ventricular hypertrophy; reperfusion injury salvage kinase
MeSH Terms: conditions — Hypertrophy, Left Ventricular | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIPC group (Experimental)
  Interventions: Procedure: Remote ischemic preconditioning at left upper arm
- Control group (Placebo Comparator)
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Remote ischemic preconditioning at left upper arm — Placement of automated cuff-inflator on the left upper arm after induction of anesthesia RIPCgroup-3 cycles of 5 min ischemia (300 mmHg inflation) & 5 min reperfusion (deflation)
  Arms: RIPC group
Procedure: Control group — keeping the cuff deflated
  Arms: Control group

SUMMARY:
The aim of this study is to investigate whether RIPC protects the heart against ischemia reperfusion injury on the concentrically hypertrophied myocardium

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥20 years with severe degenerative AS presenting concentric remodeling of the LV, who were scheduled for AVR

Exclusion Criteria:

* diabetes mellitus,
* coronary stenosis ≥70%,
* renal failure (serum creatinine > 2.0 mg/dL),
* upper arm peripheral vascular disease,
* LV ejection fraction <50%

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Serum levels of CK-MB and Tn-T | baseline
Serum levels of CK-MB and Tn-T | 12-hour after surgery
Serum levels of CK-MB and Tn-T | 24-hour after surgery

SECONDARY OUTCOMES:
Myocardial activation of protective signaling pathway | Before commencement of CPB
Myocardial activation of protective signaling pathway | After taking off CPB

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea